CLINICAL TRIAL: NCT02295826
Title: Dabigatran Following Transient Ischemic Attack and Minor Stroke
Acronym: DATAS II
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: DATAS002
Record Dates: First submitted 2014-11-17; First posted 2014-11-20 (Estimated); Last update posted 2019-01-30 (Actual); Status verified 2018-10

CONDITIONS: Transient Ischemic Attack; Minor Ischemic Stroke
MeSH Terms: conditions — Ischemic Attack, Transient | interventions — Dabigatran; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dabigatran therapy (Experimental): 150 mg BID for 30 days (dose modification - reduced to 110mg BID in patients >80 years of age and/or an eGFR of 30-50 ml/min)
  Interventions: Drug: Dabigatran
- Acetylsalicylic Acid thereapy (Active Comparator): 325 mg loading dose then 81 mg/day for 30 days
  Interventions: Drug: Acetylsalicylic acid

INTERVENTIONS:
Drug: Dabigatran — Dabigatran will be taken bid for 30 days post enrolment. The dose of dabigatran will be based on patient age and renal function.
  Other Names: Pradax (Canada)/ Pradaxa (USA and rest of world)
  Arms: Dabigatran therapy
Drug: Acetylsalicylic acid — participants randomized to ASA therapy will be loaded with 325 mg of ASA, followed by 81 mg/day
  Other Names: Aspirin
  Arms: Acetylsalicylic Acid thereapy

SUMMARY:
Rationale: To date, anticoagulant therapy in acute stroke has also been limited by excess hemorrhagic events. The oral anticoagulant dabigatran is a novel agent, which has been shown to be associated with much lower intracranial hemorrhage rates. It has been suggested that this agent may provide the superior benefits of anticoagulation in acute stroke, without the concomitant increase in hemorrhage risk associated with heparin/LMWH or warfarin.

Study Design: DATAS II is a randomized, open label blinded endpoint trial. Participants (n=300) with TIA or ischemic stroke (NIHSS score <9) will be enrolled within 48 hours of symptom onset from approximately four (4) health care centres across Canada. All participants will have an MRI with DWI lesion volume < 25 ml. Participants will be randomized 1:1 to treatment with dabigatran for 30 days or ASA 81 mg daily (current standard of care). All stroke patients will initially be screened with a non-contrast CT scan of the brain. The first MRI will be performed within 48 hours of symptom onset. Imaging studies will be repeated at day 30. All patients will be assessed clinically at Day 30 and Day 90.

Study Aims:

1. Establish the safety of early anticoagulation with the novel oral anticoagulant dabigatran in acute cerebrovascular syndrome patients.
2. Identify the rate of both symptomatic and asymptomatic hemorrhagic transformation (HT) associated with these treatments.
3. Identify predictors of HT associated with acute dabigatran treatment.

Hypothesis: The Investigators hypothesize that symptomatic HT rates in dabigatran and ASA treated patients will not be significantly different.

Study outcomes: The primary outcome is the rate of symptomatic hemorrhagic transformation (HT), defined as a parenchymal hematoma, which is >30% of the infarcted area on DWI, with substantial space- occupying effect, associated with clinical worsening (≥4 point increase in National Institutes of Health Stroke Scale (NIHSS) score) within 5 weeks of treatment initiation. The major secondary outcome the rate of asymtomatic HT see on day 30 MRI sequence.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients
2. Must be >18 years of age
3. Must have TIA or ischemic stroke (NIHSS score <9 - see section 2.7 for further clarification)
4. Symptom onset is < 72 hours prior to enrollment or Study therapy must initiated within 48 hours of symptom onset (in case where onset time cannot be established, it will be considered to be the time when the patient was lst know to be well
5. Informed consent must be obtained from either the patient or substitute decision maker (according to local REB policy) prior to any study related procedures being performed
6. All patients will have a MRI including DWI prior to randomization
7. DWI lesion volume must be <25ml
8. Patients without DWI lesions, but a clinical history considered consistent with TIA, determined by the attending physician, can be included

Exclusion Criteria:

1. Patients with stroke mimics - such as seizures, migraine etc
2. Patients with contraindications to MRI including metallic implants
3. Patients with any past sensitivity to gadolinium contrast media will be eligible, but will not undergo PWI or contrast enhanced MRA (both optional sequences)
4. Patients with renal failure defined as Glomerular Filtration Rate (GFR) < 30 ml/min
5. Patients deemed, as attending stroke physician, to have any ongoing bleeding risks or unsuitable for dabigatran therapy
6. Patients with MRI demonstrated additional pathology including arteriovenous malformations, intracranial aneurysms, tumors or abscess, which potentially increase the rise of bleed. Individuals with small incidental leasions, at low risk of bleed such as meningiomas may be included at the discretion of the investigator.
7. Patients with an acute DWI lesion volume of >25 ml (DWI volume to be estimated using the ABC/2 technique 110)**
8. Age <18 years
9. Pregnant or breast feeding women.
10. Severe dysphagia necessitating naso-gastric (NG) feeding (dabigatran can not be delivered via NG tube)
11. Planned thrombolysis or endovascular intervention for the index event
12. Thrombolysis for ischemic stroke within the preceding 7 days
13. Planned carotid endarterectomy/carotid artery stent within 30 days Note: Carotid Investigations will be completed prior to enrolment. Patients with symptomatic stenoses and a planned carotid procedure will be excluded.
14. Any history of spontaneous intracranial bleeding
15. Clear indication for anticoagulation, including atrial fibrillation, mechanical cardiac valves, deep venous thrombosis, pulmonary embolism or known hypercoagulable state
16. Co-morbid illness with expected life expectancy of <90 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2015-01; Primary Completion 2018-12-18 (Actual); Study Completion 2018-12-18 (Actual)

PRIMARY OUTCOMES:
Rate of symptomatic hemorrhagic transformation | within 5 weeks of treatment initiation
  The primary endpoint is the rate of symptomatic hemorrhagic transformation (HT), defined as a parenchymal hematoma, which is >30% of the infarcted area on DWI, with substantial space-occupying effect, associated with clinical worsening (≥4 point increase in National Institutes of Health Stroke Scale (NIHSS) score) within 5 weeks of treatment initiation.

SECONDARY OUTCOMES:
Rate of asymtomatic hemorrhagic transformation | day 30

CONTACTS AND LOCATIONS:
Locations (6):
- Canada (6):
  - University of Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - Grey Nuns Hospital, Edmonton, Alberta
  - Vancouver Stroke Program, Vancouver, British Columbia
  - Hamilton Health Sciences, Hamilton, Ontario
  - Centre Hospitalier de l'Université de Montréal, Hôpital Notre-Dame, Montreal, Quebec

REFERENCES:
- [Derived] Cimen E, Ng K, Buck BH, Field T, Coutts SB, Gioia LC, Hill MD, Miller J, Benavente OR, Sharma M, Butcher K. Importance of infarct topography in determination of stroke mechanism and recurrence risk: a post-hoc analysis of the dabigatran acute treatment of stroke trial. BMJ Open. 2025 Jan 9;15(1):e087704. doi: 10.1136/bmjopen-2024-087704. PMID 39788764
- [Derived] Alrohimi A, Rose DZ, Burgin WS, Renati S, Hilker NC, Deng W, Oliveira GH, Beckie TM, Labovitz AJ, Fradley MG, Tran N, Gioia LC, Kate M, Ng K, Dowlatshahi D, Field TS, Coutts SB, Siddiqui M, Hill MD, Miller J, Jickling G, Shuaib A, Buck B, Sharma M, Butcher KS. Risk of hemorrhagic transformation with early use of direct oral anticoagulants after acute ischemic stroke: A pooled analysis of prospective studies and randomized trials. Int J Stroke. 2023 Aug;18(7):864-872. doi: 10.1177/17474930231164891. Epub 2023 Mar 26. PMID 36907985
- [Derived] Butcher KS, Ng K, Sheridan P, Field TS, Coutts SB, Siddiqui M, Gioia LC, Buck B, Hill MD, Miller J, Klahr AC, Sivakumar L, Benavente OR, Hart RG, Sharma M. Dabigatran Treatment of Acute Noncardioembolic Ischemic Stroke. Stroke. 2020 Apr;51(4):1190-1198. doi: 10.1161/STROKEAHA.119.027569. Epub 2020 Feb 26. PMID 32098609
- [Derived] Ng KH, Sharma M, Benavente O, Gioia L, Field TS, Hill MD, Coutts SB, Butcher K; DATAS-2 Investigators. Dabigatran following acute transient ischemic attack and minor stroke II (DATAS II). Int J Stroke. 2017 Oct;12(8):910-914. doi: 10.1177/1747493017711947. Epub 2017 Jun 6. PMID 28585903